CLINICAL TRIAL: NCT05820243
Title: Determinants of Changes in Arterial Load Following Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, David Edwards, Professor, University of Delaware
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1783804
Record Dates: First submitted 2023-03-16; First posted 2023-04-19 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Post-Exercise Hypotension
Keywords: arterial stiffness; wave reflections; pulsatile load
MeSH Terms: conditions — Post-Exercise Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Antihistamine and placebo treatments will be provided in opaque gel capsules by a member of the research team not involved in data collection or analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antihistamine (Experimental): The oral antihistamine condition will consist of fexofenadine (540mg) and famotidine (40mg). Commercially available pills (3 x 180mg fexofenadine and 2 x 20mg famotidine) will be placed within opaque capsules and administered to the participants upon arrival to the laboratory.
  Interventions: Other: Moderate Intensity Aerobic Exercise
- Placebo (Placebo Comparator): The placebo condition will consist of dextrose in an identical number of opaque capsules as the antihistamine treatment. Total dextrose will be <5g. The capsules will be administered to the participants upon arrival to the laboratory.
  Interventions: Other: Moderate Intensity Aerobic Exercise

INTERVENTIONS:
Other: Moderate Intensity Aerobic Exercise — Participants will complete 1 hour of exercise on a cycle ergometer at the power output that elicits 60% of their peak rate of oxygen consumption (V02peak).

SUMMARY:
The goal of this study is to learn about how blood vessel dilation after exercise effects pulse wave reflection and influences the function of the heart in healthy young adults. The main question it aims to answer is: Are post-exercise decreases in reflected pulse waves due to a decrease in the stiffness of large arteries in the leg or an increase in leg blood flow? Participants will exercise on a stationary bicycle at a moderate intensity for 1 hour during two laboratory visits. Participants will take oral antihistamines to block post-exercise dilation at one visit, and they will take placebo pills at the other visit. At both visits, leg blood flow, pulse wave velocity, and heart function will be measured before exercise and for 120-minutes after exercise.

DETAILED DESCRIPTION:
During exercise, blood vessels increase in size to supply muscles with more blood. After exercise, the muscles that had been used release chemicals called histamines that cause the blood vessels to stay dilated even when the muscles no longer need more blood. It takes around 2 hours for the blood vessels to return to normal. This causes blood pressure to be lower than it usually is at rest. This phenomenon delays the return of pressure waves in arteries that are reflected back to the heart resulting in the heart having to work less hard to pump out blood for about 2 hours after exercise. However, it is unknown why the reflected pressure waves return to the heart later. The aim of this study is to determine if this delay is due to the speed of the reflected waves being slowed by large arteries or dilation of small arteries resulting in the reflections originating further from the heart. By giving antihistamines prior to exercise, post-exercise blood vessel dilation of the small arteries will be largely reduced, thus allowing for the determination of which factor causes the reflected waves to return later. Additionally, it is hypothesized that the reduction in work that the heart must perform results in improved contraction and relaxation of the heart. Thus, an additional aim is to determine how post-exercise blood vessel dilation influence heart function.

To accomplish these aims, blood flow leaving the left ventricle and femoral blood flow will be measured via Doppler ultrasound. Applanation tonometry will be used to record pulse waves at the carotid, radial, femoral, and dorsalis pedis arteries. These pulse waves will be used to estimate central blood pressure and to determine pulse wave velocity of different arterial segments. Measurements will be made at baseline and for 120 minutes after a bout of moderate intensity aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* sedentary or recreationally active

Exclusion Criteria:

* history of cardiovascular events or procedures
* stage 2 hypertension (BP: ≥140 systolic or ≥90 diastolic)
* metabolic syndrome
* renal disease
* chronic respiratory disease
* currently prescribed any cardiovascular medication
* current use of erythromycin and/ ketoconazole
* current pregnancy or breastfeeding -hormone replacement therapy-
* tobacco use
* musculoskeletal injury/disorder that would inhibit cycling exercise
* body mass index (BMI) <18.5 or >35kg/m^2
* reduced kidney function (estimated glomerular filtration rate< 90ml/min/1.73 m^2)
* daily use of fexofenadine and/or famotidine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in lower limb arterial stiffness | 120 minutes post-exercise
  Arterial stiffness of the leg will be assessed via measurement of femoral-pedis pulse wave velocity.
Change in leg vascular conductance | 120 minutes post-exercise
  Vascular conductance, an index of peripheral vasodilation, will be determined by measuring femoral blood flow via ultrasound and dividing by mean arterial pressure.
Change in left ventricular pulsatile load | 120 post-exercise
  Doppler echocardiography and arterial tonometry will be used to establish left ventricular pressure-flow relations. Wave separation analysis will subsequently be performed to determine the magnitude and timing of reflected pulse waves.

SECONDARY OUTCOMES:
Change in left ventricular diastolic function | 120 minutes post-exercise
  Echocardiographic measures of left ventricular diastolic function will be recorded, including mitral annulus tissue velocity and mitral in-flow velocity

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Kinesiology and Applied Physiology, University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided